CLINICAL TRIAL: NCT02980120
Title: Personality Pathology and Cerebral Processing in Eating Disorders
Acronym: EAT_FMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Kathrin Sevecke, Univ.-Prof. Dr. med., Medical University Innsbruck
Other Study IDs: EAT_FMRI
Record Dates: First submitted 2016-11-09; First posted 2016-12-02 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa | interventions — Wechsler Scales; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Anorexia Nervosa Group: n=50 female patients with Anorexia Nervosa (AN) who fulfill the criteria for DSM-IV, BMI z-scores will be used for age and sex specific cut-off points that are extrapolated from the adult BMI cut-off <17.5 Interventions:EDI-2, EAT, SCID-I, SCID-II, LoPF, HAWIK-IV, fMRI
  Interventions: Other: SCID-I; Other: EAT; Other: EDI-2; Other: SCID-II; Other: LoPF; Other: HAWIK-IV; Device: fMRI
- Bulimia Nervosa Group: n=30 female patients with Bulimia Nervosa (BN) who have BMI z-scores from the adult range <17.5-25.0 (this reflects the lower prevalence rates of BN compared to AN) Interventions:EDI-2, EAT, SCID-I, SCID-II, LoPF, HAWIK-IV, fMRI
  Interventions: Other: SCID-I; Other: EAT; Other: EDI-2; Other: SCID-II; Other: LoPF; Other: HAWIK-IV; Device: fMRI
- Healthy Control Group: n=30 healthy females who have BMI z-scores from the adult range from 19.0-25.0 and who do not fulfill diagnostic criteria for any psychiatric disorder.Interventions:EDI-2, EAT, SCID-I, SCID-II, LoPF, HAWIK-IV, fMRI
  Interventions: Other: SCID-I; Other: EAT; Other: EDI-2; Other: SCID-II; Other: LoPF; Other: HAWIK-IV; Device: fMRI

INTERVENTIONS:
Other: SCID-I — The structured clinical interview for DSM-IV Axis I Disorder (SCID-I, German translation, see Wittchen, Zaudig & Fydrich, 1997) is a semi-structured interview to diagnose AN and BM. It allows a detailed assessment of ED symptoms across different settings and time periods necessary to make an accurate diagnosis.
  Other Names: Structured Clinical Interview for DSM-IV
Other: EAT — The Eating Attitudes Test (EAT) is a standardized questionnaire of symptoms and concerns related to ED (Garner & Garfield, 1979, German translation by Steinhausen). The questionnaire consists of 40 items on a six-point Likert scale, providing information
  Other Names: Eating Attitudes Test
Other: EDI-2 — The Eating Disorder Inventory 2 (Paul & Thiel, 2004) is a self-report questionnaire on psychological features generally associated with AN and BN.The instrument consists of 91 items on a six-point Likert scale. The 11 scales are drive for thinness, bulimia, body dissatisfaction, ineffectiveness, perfectionism, interpersonal distrust, interoceptive awareness, maturity fears, asceticism (provisional), impulse regulation (provisional) and social insecurity (provisional). It was designed as a diagnostic aid; its psychometrics have been tested, with studies demonstrating satisfactory internal consistency reliability coefficients (between .44 and .93), test-retest reliability of .79 to .95 (after one week) and above .80 (after three weeks), and content, convergent and discriminant validity.
  Other Names: Eating Disorder Inventory 2
Other: SCID-II — The SCID-II interview (German, see Wittchen, Zaudig & Fydrich, 1997) is a widely used and researched instrument to assess DSM-IV-TR personality disorders.The interview covers all ten DSM-IV personality disorders (antisocial, avoidant, borderline, dependent, histrionic, narcissistic, obsessive-compulsive, paranoid, schizoid and schizotypal), PD not otherwise specified, and appendix categories (depressive PD and passive-aggressive PD) and is used to make personality disorder diagnoses either dimensionally or categorically (present-absent). Furthermore, it allows the investigation of patterns of PD that co-occur with other mental disorders as well as the analysis of the underlying structure of personality pathology.
  Other Names: Structured Clinical Interview for DSM-IV
Other: LoPF — In order to specifically focus on certain personality traits, we use the LoPF as an additional measure. It is a well-validated and reliable self-report questionnaire to measure healthy and pathological personality functioning in adolescents. It is based on the DSM-5 Section III Alternative Model for Personality disorders and covers core impairments in adolescents' personality functioning: identity, self-direction (self-related personality functioning), intimacy/ attachment and empathy/ social-related personality functioning (Sevecke & Krischer, 2011).
  Other Names: Levels of personality functioning
Other: HAWIK-IV — The Wechsler Intelligence Scale for Children (HAWIK-IV, Petermann & Petermann, 2008) will be used assess intelligence. For adolescents older than 16.11 years, we will use the German version of the Wechsler Adult Intelligence Scale (HAWIE-IV).Results from test-retest reliability demonstrate that the mean retest scores for all subtests are higher than the mean test scores from first administration, with effect sizes ranging from .08 (comprehension) to .60 (picture completion). The test has demonstrated an acceptable relationship to other measures of achievement, memory, adaptive behavior, emotional intelligence and giftedness in children and adolescents (Canivez, 2014). For the non-clinical adolescent sample, we will use two subtests of the HAWIK.
  Other Names: Wechsler Intelligence Scale for Children
Device: fMRI — To measure food-related brain activation, event-related fMRI will be used, with phases of high-caloric images alternating with phases of low-caloric images and images of fixation cross (not related to food images). A total of 18 blocks will be performed - see figure below. The duration of each phase will be 30 seconds. In a second run, the patients and control subjects will drink chocolate milk and water, alternating every 30 seconds, through a long silicon tube. This procedure was successfully tested in a previous fMRI study with adult AN patients (Gizewski et al. 2010, Vocks et al. 2011) and has now been adopted in preliminary measurements for young AN patients.
  Other Names: Food-related brain activation by event-related fMRI

SUMMARY:
The proposed study will investigate whether, on the basis of personality traits and personality disorders as well as specific cerebral activation patterns shows differences in adolescent female with anorexia nervosa (AN), bulimia nervosa (BN) and a healthy control group.

DETAILED DESCRIPTION:
The increasing prevalence of eating disorders in adolescence and their frequent chronic course have led to the development of various programs for prevention, early detection and early intervention. Nevertheless, the causes of anorexia nervosa (AN) and bulimia nervosa (BN) remain a topic of much discussion and research. Evidence points to a multifactorial disease pattern in which intrapsychic, psychosocial and biological factors interact and reinforce one another. Eating disorders have been increasingly associated with signs of emotional and psychological disturbance. In clinical populations, personality traits are observed as exacerbating factors that constitute important variables for differentiation. While investigations have shown high comorbidity of personality disorders and eating disorders in adulthood, comparable studies in adolescence have not yet been undertaken.

The proposed study will investigate whether, on the basis of personality traits and personality disorders as well as specific cerebral activation patterns, differentiations can be identified among adolescent female patients with AN (n = 50) and BN (n = 30) in comparison to a healthy control group (n = 30).

Of particular interest is the potential connection between specific personality traits and neural correlates in the two ED:

1. Do specific personality traits and personality disorders correlate significantly with particular types of ED?
2. Do AN and BN correlate significantly with particular cerebral activation patterns following visual presentation of food stimuli and gustatory stimuli? 3. Can connections be identified between specific personality profiles and cerebral activation patterns in AN and BN? 4. Will changes in cerebral activation patterns be evident between the beginning of treatment (T1) and the end of treatment (T2)? The study will use specific questionnaires dealing with eating behavior (EDI & EAT) as well as clinical interviews for the assessment of personality disorders (SCID II). Cerebral processing will be evaluated using functional MRI (fMRI) and structural MRI. fMRI results from visual and gustatory stimuli will be correlated with structural brain morphology in MRI and with psychopathological parameters. The correlation of such clinical values represents a new approach to the investigation of eating disorders in adults and may be of significant relevance for data interpretation and understanding of cerebral changes due to anorexia. MRI measurements will be performed at begin of therapy (T1) and at end of therapy (T2).

In this fashion, known risk factors will be supplemented with information on specific personality traits and cerebral activation patterns. The proposed study will thus provide important new insights for early detection, prevention, treatment and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

• The study will include 50 female patients with AN, 30 female patients with BN and 30 healthy females

Exclusion Criteria:

* Age >18 years or <14 years
* Extremely underweight patients requiring pediatric treatment for medical stability and improvement of cognitive functioning prior to psychiatric inpatient treatment Overweight and obese patients with BMI z-scores extrapolated from the adult BMI cut-off > 25.0
* Acute or chronic somatic or functional diseases (i.e. strokes, tumors, heart conditions)
* A history of head trauma or fainting
* Left-handedness (determined by a standardized questionnaire)
* Evidence of structural brain abnormality on the structural MRI scan (conducted on the first day of the study)
* fMRI-specific exclusion criteria (phobic anxiety, claustrophobia, ADHD etc.)
* Pregnancy (assessed with urine pregnancy test)
* Allergy to chocolate
* Schizophrenia and other psychotic disorders
* Shrapnel or other electronic/metal implants in the body (i.e. pacemakers, surgical devices etc.)

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include 50 female patients with AN, 30 female patients with BN and 30 healthy females
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Neural correlates (fMRI): Differences on cerebral activation patterns in the AN and BN groups from those in the control group | At the begin of therapy (T1, week 1) and at the end of therapy (T2) (approx. 2 months)
  Cerebral activation patterns ((activation of prefrontal, parahippocampal, cinculate, and insular cortex, posterior cingulate cortex ) in the AN and BN groups will differ from those in the control group

SECONDARY OUTCOMES:
Personality pathology: Identification of specific personality profiles (dimensional personality traits and personality disorders) using a structured clinical interview and questionnaire | (T1) Week 1
  Specific personality profiles (dimensional traits and personality disorders) can be identified in adolescent patients with AN and BN; evaluated from SCID-II interview (scores ranging from 108-324) and LoPF questionnaire (T-scores)
Relationship between personality pathology (using structured clinical interview and questionnaire) and neural correlates in ED (fMRI) | At the begin of therapy (T1, week 1) and at the end of therapy (T2) (approx. 2 months)
  Personality pathology will correlate significantly with the cerebral activation patterns (fMRI brain activation, SCID-scores and T-scores)

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Seveke, Univ-Prof.Dr, Principal Investigator — Head of department of Child and Adolescent Psychiatry
Locations (1):
- Department for Child and Adolescent Psychiatry, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dabkowska-Mika A, Steiger R, Gander M, Haid-Stecher N, Fuchs M, Sevecke K, Gizewski ER. Evaluation of visual food stimuli paradigms on healthy adolescents for future use in fMRI studies in anorexia nervosa. J Eat Disord. 2023 Mar 6;11(1):35. doi: 10.1186/s40337-023-00761-8. PMID 36879292